CLINICAL TRIAL: NCT01785589
Title: Stress Thallium-201/Rest Technetium-99m Sequential Dual Isotope High-Speed Myocardial Perfusion Imaging Validation Versus Invasive Coronary Angiography
Brief Title: Validation of Myocardial Perfusion Imaging
Acronym: CameraCZT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IRB 5891
Record Dates: First submitted 2013-01-29; First posted 2013-02-07 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; cardiac nuclear medicine; myocardial perfusion imaging; invasive coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- coronary angiography-FFR-CZT (Other): Patients who were referred to our cardiology department for stress-rest CZT SPECT for known or suspected CAD and submitted for a clinical reason to invasive coronary angiography within 2 month of the SPECT studies. for these patients, A 6 French arterial sheath was introduced into the radial artery. After administration of 5000 U heparin, the guiding catheter was advanced into the coronary ostium. Intracoronary nitroglycerin 0.2 mg was administered, and reference images were made. Significant CAD was defined as presentation of a stenosis ≥70 % in the three-epicardial vessels and ≥ 50 % in left main coronary disease. If necessary (at the discretion of the practitioner) the pressure wire was advanced across the stenosis, and Fractional flow reserve (FFR) was measured.
  Interventions: Procedure: coronary angiography

INTERVENTIONS:
Procedure: coronary angiography — A 6 French arterial sheath was introduced into the radial artery. After administration of 5000 U heparin, the guiding catheter was advanced into the coronary ostium. Intracoronary nitroglycerin 0.2 mg was administered, and reference images were made. Significant CAD was defined as presentation of a stenosis ≥70 % in the three-epicardial vessels and ≥ 50 % in left main coronary disease. If necessary (at the discretion of the practitioner) the pressure wire was advanced across the stenosis, and Fractional flow reserve (FFR) was measured.
  Other Names: Coronary angiography = using standard techniques (Philips Allura Xper FD10, Philips Healthcare); Pressure wire = Certus; St. Jude Medical, St. Paul, Minnesota; FFR by using RadiAnalyzer =St. Jude Medical, St. Paul, Minnesota); intravenous adenosine = ADENOSCAN 30mg/10ml S perf IV 6Fl/10ml (Sanofi-Aventis France)

SUMMARY:
The new cadmium-zinc-telluride (CZT) technology is a powerful tool for cardiac nuclear medicine. The increased photon counting sensitivity of camera can be used to explore novel protocols like dual isotope (rapid stress Tl-201/rest Tc-99m protocol for use with high-speed SPECT MPI). The use of dual isotope imaging is very interesting because this imaging combines the use of thallium-201 with technetium-99m agents permitting optimal image resolution and simultaneous assessment of viability, all with an exam duration of approximately 20 minutes. However, no study compares stress thallium-201/rest technetium-99m sequential dual isotope high-speed myocardial perfusion imaging versus invasive coronary angiography. The investigators report here the first validation of high-speed protocol with dual isotope for myocardial perfusion imaging using invasive coronary angiography as the standard of reference.

DETAILED DESCRIPTION:
The new cadmium-zinc-telluride (CZT) technology is a powerful tool for cardiac nuclear medicine. Indeed, recent clinical validation studies of CZT technology have documented a scan time reduction and low radiation dose without degradation of myocardial perfusion imaging in comparison with standard dual detector cameras. The increased photon counting sensitivity of camera can be used to explore novel protocols that may offer advantages over standard protocols used for Myocardial Perfusion Imaging. Berman et al. showed that rapid stress Tl-201/rest Tc-99m protocol for use with high-speed SPECT MPI has offered the superior qualities of Tl-201 for stress imaging and of the Tc-99m agents for rest imaging can be preserved. Nuclear medicine presents the most level of scientific validation for diagnosis and prognosis of coronary artery disease. A lot of studies have compared performance of standard dual detector cameras vs. Invasive Coronary Angiography. Fiechter et al. reported the first validation of ultrafast dedicated cardiac gamma camera with CZT versus invasive coronary angiography. But he used a novel hybrid SPECT /CT device and 99m-Tc-tetrofosmin pharmacological stress/rest examination. However, no study compares stress thallium-201/rest technetium-99m sequential dual isotope high-speed myocardial perfusion imaging versus invasive coronary angiography. Moreover, diagnosis performance of this high-speed protocol versus fractional flow reserve for stenosis evaluation is unknown.

The investigators report here the first validation of high-speed protocol with dual isotope for myocardial perfusion imaging using invasive procedures (coronary angiography and fractional flow reserve) as the standard of reference.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina
* Cadmium-zinc-telluride gamma camera SPECT with dual isotope imaging
* Coronarography

Exclusion Criteria:

* Pregnant woman
* Patient with terminal illness,
* Terminal Renal failure
* Allergy to iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Accuracy, positive and negative predictive value of Stress Thallium-201/Rest Technetium-99m Sequential Dual Isotope High-Speed Myocardial Perfusion Imaging to detect coronary artery disease | 2 months
  Diagnostic performance of Stress Thallium-201/Rest Technetium-99m Sequential Dual Isotope High-Speed Myocardial Perfusion Imaging to detect coronary artery disease is evaluated vs. coronary angiography.
  Significant CAD was defined as presentation of a stenosis ≥70 % in the three-epicardial vessels and ≥ 50 % in left main coronary disease in coronary angiography.
  In CZT SPECT, The global summed stress score (SSS) summed rest score (SRS) and summed difference score (SDS) were calculated by adding the scores of the 17 segments in the stress and rest images, respectively. Significant ischemia is defined by SSS >4.
  Analyze is performed per patients, per segments, and per vessels.

SECONDARY OUTCOMES:
Accuracy, positive and negative predictive value of Stress Thallium-201/Rest Technetium-99m Sequential Dual Isotope High-Speed Myocardial Perfusion Imaging to detect coronary artery disease | 2 months
  Diagnostic performance of Stress Thallium-201/Rest Technetium-99m Sequential Dual Isotope High-Speed Myocardial Perfusion Imaging to detect coronary artery disease is evaluated vs. Fractional Flow reserve (FFR).
  Significant CAD was defined as presentation of a stenosis with FFR ≤ 0.8 in the three-epicardial vessels and in left main coronary disease.
  In CZT SPECT, The global summed stress score (SSS) summed rest score (SRS) and summed difference score (SDS) were calculated by adding the scores of the 17 segments in the stress and rest images, respectively. Significant ischemia is defined by SSS >4.
  Analyze is performed per patients, per segments, and per vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles GB Barone-Rochette, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France

REFERENCES:
- [Derived] Barone-Rochette G, Leclere M, Calizzano A, Vautrin E, Celine GC, Broisat A, Ghezzi C, Baguet JP, Machecourt J, Vanzetto G, Fagret D. Stress thallium-201/rest technetium-99m sequential dual-isotope high-speed myocardial perfusion imaging validation versus invasive coronary angiography. J Nucl Cardiol. 2015 Jun;22(3):513-22. doi: 10.1007/s12350-014-0016-0. Epub 2014 Nov 8. PMID 25381092